CLINICAL TRIAL: NCT02665208
Title: Mobile Phone Messaging to Support Smoking Cessation Among Office-based Buprenorphine and Inpatient Detoxification Patients: a Pilot Study
Brief Title: A Pilot Text Messaging Intervention to Reduce Smoking in Office-based Buprenorphine and Inpatient Detoxification Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-01654
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Smoking Cessation
Keywords: cigarettes; smoking; opiate-dependence; alcohol; detoxification
MeSH Terms: conditions — Smoking Cessation; Smoking; Opioid-Related Disorders | interventions — Therapeutics; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment As Usual (TAU) (Active Comparator): Participants will receive informational pamphlets and information for a 1800 quit line, and a prescription for a nicotine replacement therapy (NRT) for 7 Days
  Interventions: Other: Treatment As Usual (TAU)
- Nicotine Replacement Therapies (Active Comparator): Participants will receive a prescription for a nicotine replacement therapy (NRT) for 7 Days.
  Interventions: Drug: Nicotine Replacement Therapies
- Text Message Intervention (Active Comparator): Participants will receive up to 5 messages a day with message content informed by principles of cognitive behavioral therapy using software developed and maintained by the National Cancer Institute.
  Interventions: Behavioral: Text Message Intervention (TMI)

INTERVENTIONS:
Other: Treatment As Usual (TAU) — informational pamphlets and information from 1800 quit line + prescription for nicotine replacement therapy (NRT) based on on the quantity of baseline self-reported smoking, or nicotine replacement gum (2mg)
  Arms: Treatment As Usual (TAU)
Drug: Nicotine Replacement Therapies — a prescription for a nicotine replacement therapy (NRT) (i.e. nicotine replacement patches based on the quantity of baseline self-reported smoking, or nicotine replacement gum (2mg)
  Arms: Nicotine Replacement Therapies
Behavioral: Text Message Intervention (TMI)
  Arms: Text Message Intervention

SUMMARY:
The primary purpose of this study is to understand the feasibility of a text messaging intervention developed by the National Cancer Institute, known as Smokefreetxt, to improve smoking cessation among opiate and/or alcohol dependent participants discharged from an inpatient detoxification unit and enrolled in an office-based buprenorphine program patients (OBBP). Participants will be randomized to 1) treatment as usual (TAU) comprised of informational pamphlets and information for a 1800 quit line; and a prescription for a nicotine replacement therapy (NRT) (i.e. nicotine replacement patches based on the quantity of baseline self-reported smoking, or nicotine replacement gum (2mg) #10, for 28 days which is offered routinely to all inpatients at Bellevue at the time of discharge) versus the SmokeFreeTXT intervention plus prescriptions for NRT.

ELIGIBILITY:
Inclusion Criteria:

* self-described every or some day smoker
* diagnosed with opiate dependence and/or alcohol dependence (DSM-IV) per Physician medical records (MISYS)
* Fluency in English and able to provide a written informed consent
* Currently owning a mobile phone with a working phone number
* Expected to reside in the New York City area for the next 12 months
* Understands and able to respond to the intervention text message

Exclusion Criteria:

* inability to read or understand English
* currently using nicotine replacement therapies (patch, gum, e-cigarettes), pharmacotherapy for smoking cessation such as bupropion (zyban, wellbutrin), varenicline (Chantix).
* suicidal or homicidal ideations
* any ongoing psychotic disorder, life-threatening medical or psychiatric condition
* leaves the inpatient detoxification unit prior to completing study enrollment
* is pregnant, nursing or planning to conceive within the duration of the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Difference in patient acceptability assessed via rates of participant adoption of TMI | 24 Weeks
Feasibility measured by rates of retention in the TMI | 24 Weeks
Clinical impact assessed using self-reported abstinence at week 1 via a text message inquiry from study | 24 Weeks

SECONDARY OUTCOMES:
Change in pattern of mobile device, computer, and internet usage. | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Babak Tofighi, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States